CLINICAL TRIAL: NCT03796455
Title: Effects of Low Dose of Fish Oil (EPA+DHA) vs. Combined EPA+DHA and HMB Supplementation on Protein Metabolism, Muscle Mass and Functional Capacity in Moderate to Severe COPD
Brief Title: Fish Oil and HMB Supplementation in COPD
Acronym: COPD fish oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0870
Record Dates: First submitted 2018-09-28; First posted 2019-01-08 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Fish Oil supplement; HMB supplement
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fish Oil (Experimental): 2.0 g EPA + DHA / day + placebo powder
  Interventions: Dietary Supplement: Capsule + Powder supplementation; Other: stable tracer infusion
- Fish Oil and HMB (Experimental): 2.0 g EPA + DHA + 3.0 g HMB / day
  Interventions: Dietary Supplement: Capsule + Powder supplementation; Other: stable tracer infusion
- Placebo (Placebo Comparator): 3 g/d soy oil: corn oil (50:50 ratio) + placebo powder
  Interventions: Dietary Supplement: Capsule + Powder supplementation; Other: stable tracer infusion

INTERVENTIONS:
Dietary Supplement: Capsule + Powder supplementation — For Fish oil and Placebo oil, treatment will be provided in capsules.Each group will receive dose distributed to 3 capsules per day. Participants will be instructed to take all capsules with morning meal. . For HMB and a placebo powder, product will be delivered as powder taken with water or non-carbonated beverage (like juice). Product will be provided in 2 sachets/day. One sachet should be consumed with breakfast and the other prior to bedtime (approx. 10pm).
Other: stable tracer infusion — labeled amino acids L-Phenylalanine (ring-13C6), L-Tyrosine (ring-D4), and tau-Methylhistidine will be infused as a single injection. Subsequently, the catheter will be used for arterialized venous blood samples (3 ml) drawn multiple through the day

SUMMARY:
In the present study, the role of chronic (10 weeks) intake of low dose (2g/day) of EPA+DHA in whole body protein metabolism, and functional performance and systemic inflammation will be examined, and whether adding either HMB at 3.0 g/d to the low dose of EPA+DHA (2.0 g/d) will enhance these effects even more.

DETAILED DESCRIPTION:
Weight loss commonly occurs in patients with Chronic Obstructive Pulmonary Disease (COPD), negatively influencing their quality of life, treatment response and survival. Furthermore, limb muscle dysfunction (weakness and/or enhanced fatigue) is a major systemic comorbidity in patients with Chronic Obstructive Pulmonary Disease (COPD), negatively affecting their exercise performance, physical activity, quality of life, and mortality. As nutritional abnormalities are main contributors to muscle loss and dysfunction in COPD, nutritional support is viewed as an essential component of integrated care in these patients.

Although nutritional support is effective in the treatment of weight loss in COPD, attempts to increase muscle mass and function in COPD by supplying large amounts of protein or calories to these patients have been small. This suggests that gains in muscle mass and function are difficult to achieve in COPD unless specific metabolic abnormalities are targeted. The investigators and other researchers found that low muscle mass in COPD was strongly associated with elevated whole body protein turnover and increased myofibrillar protein breakdown rates indicative of muscle contractile protein loss. The investigators have extended this finding recently to normal weight COPD patients characterized by muscle weakness using a more precise and accurate pulse method of tau-methylhistidine tracer.

A substantial number of COPD patients, underweight as well as normal weight to obese, are characterized by an increased inflammatory response as evidenced by elevated levels of the pro-inflammatory cytokines (Tumor Necrosis Factor (TNF)-α, Interleukin (IL) 6 and 8, and the soluble TNF-α receptors (55 and 75). Furthermore, CRP levels are elevated in COPD and associated with reduced quadriceps strength, lower maximal and submaximal exercise capacity and increased morbidity.

One of the few agents capable to suppress the generation of pro-inflammatory cytokines are eicosapentanoic acid (EPA) and docosahexanoic acid (DHA), primary ω-3 fatty acids found in fish oils.

Previous experimental research and clinical studies in cachectic conditions (mostly malignancy) indicate that polyunsaturated fatty acids (PUFA) are able to attenuate protein degradation by improving the anabolic response to feeding and by decreasing the acute phase response. Eicosapentaenoic acid (EPA), in combination with docosahexaenoic acid (DHA), has been shown to effectively inhibit weight loss in several disease states, however weight weight and muscle mass and function increase was not present or minimal. Also in healthy older adults, fish oil can slow the decline in muscle mass and function. A randomized clinical trial in COPD patients showed that extra nutritional supplementation with PUFAs daily of 1000 mg EPA+DHA as adjunct to exercise training during 8 weeks enhanced exercise capacity but did not lead to muscle mass gain. The patients who did not respond adequately (< 2% gain in weight), had a higher TNF-α level than those who did gain sufficient weight, which is in line with previous data in COPD showing an association between an increased systemic inflammation with non-response to nutritional therapy.

Although previous studies support the concept of EPA+DHA supplementation to ameliorate the systemic inflammatory response and decrease protein breakdown, there is no information present on the effects of EPA+DHA supplementation on whole body and muscle protein metabolism in COPD. The investigators have recently examined the dose-response effects of 0, 2 and 3.5 g of EPA+DHA intervention ( EPA / DHA) for 4 weeks in stable moderate to severe COPD patients (8pts /group) (unpublished data) but were not able to find a positive effect of muscle mass and strength, even with the highest dose, likely related to the relatively short (4 week) supplementation period. The effect of EPA+DHA intervention on whole body and muscle protein synthesis and breakdown rates is currently being analysed.

Although numerous animal studies have shown the benefit of HMB in downregulating muscle protein breakdown under catabolic conditions, there is very little data in COPD patients. Others have tested HMB (3g/d) in COPD patients in the ICU and reported anti-inflammatory benefits and improvement in pulmonary function. In patients with bronchiectasis, 24 week supplementation with an ONS containing HMB (1.5g/d) versus standard of care during pulmonary rehabilitation program, resulted in benefits on body composition, muscle strength and QoL. A combination of HMB and EPA/DHA in a mouse model of cancer cachexia showed a synergy between the two ingredients on preventing muscle loss and downregulation of muscle protein degradation.

ELIGIBILITY:
Inclusion criteria

* Ability to walk, sit down and stand up independently
* Ability to lie in supine or slightly elevated position for 8.5 hours
* Age 45 - 100
* Clinical diagnosis of COPD, including moderate to very severe chronic airflow limitation, and an FEV1 < 70% of reference FEV1 (GOLD II-III). If subjects are on β2 agonists, only those subjects with <10% improvement in FEV1 will be included.
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol, including:

  * Refraining from intense physical activities (72h) prior to each study visit
  * Adhering to fasting state and no smoking from 10 pm ± 2h onwards the day prior to each study visit

Exclusion Criteria

* Participants 86 and older that fail to get physician approval
* Established diagnosis of malignancy
* Established diagnosis of Insulin Dependent Diabetes Mellitus
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* BMI ≥ 45 kg/m2
* Dietary or lifestyle characteristics:

  * Daily use of supplements containing EPA+DHA or HMB prior to the first test day
  * Use of protein or amino acid containing nutritional supplements within 5 days of first test day
  * Indications related to interaction with study products. Known hypersensitivity to fish and/or shellfish and/or soy
  * Use of long-term oral corticosteroids or short course of oral corticosteroids 4 weeks preceding first test day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Changes to net whole body protein metabolism | baseline and after 10-week supplementation
  whole body protein synthesis and myofibrillar protein breakdown measured by labeled amino acids on each study day via blood drawn at time 4, 10, 15, 20, 30, 40, 60, 120, 180, 240 minutes of infusion

SECONDARY OUTCOMES:
muscle mass | 15 minutes on baseline visit, visit at week 5 of supplement intake, and after 10-week supplementation
  Body composition as measured by Dual-Energy X-ray Absorptiometry
limb muscle strength | 15 minutes on baseline visit, visit at week 5 of supplement intake, and after 10-week supplementation
  kin-com 1-leg test
respiratory muscle strength | 15 minutes on baseline visit, visit at week 5 of supplement intake, and after 10-week supplementation
  Micro-respiratory pressure meter to measure maximum inspiratory and expiratory pressure
functional performance via six minute walk test | baseline visit, visit at week 5 of supplement intake, and after 10-week supplementation
  walk a predetermined loop of 69.77 meters (228.89 feet) at self-selected pace for six minutes
systemic inflammatory markers | baseline visit and after 10-week supplementation
  blood sample will be taken to measure c-reactive protein levels
resting energy expenditure | baseline visit and after 10-week supplementation
  Oxygen consumption and carbon dioxide production will be calculated from the airflow in a transparent plastic (Plexiglas) hood to determine concentration differences between inhaled and exhaled air

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelen MPKJ, Simbo SY, Ruebush LE, Thaden JJ, Ten Have GAM, Harrykissoon RI, Zachria AJ, Calder PC, Pereira SL, Deutz NEP. Functional and metabolic effects of omega-3 polyunsaturated fatty acid supplementation and the role of beta-hydroxy-beta-methylbutyrate addition in chronic obstructive pulmonary disease: A randomized clinical trial. Clin Nutr. 2024 Sep;43(9):2263-2278. doi: 10.1016/j.clnu.2024.08.004. Epub 2024 Aug 10. PMID 39181037
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Pinson MR, Deutz NEP, Harrykissoon R, Zachria AJ, Engelen MPKJ. Disturbances in branched-chain amino acid profile and poor daily functioning in mildly depressed chronic obstructive pulmonary disease patients. BMC Pulm Med. 2021 Nov 7;21(1):351. doi: 10.1186/s12890-021-01719-9. PMID 34743729